CLINICAL TRIAL: NCT02959034
Title: Pediatric Metabolism and Microbiome Repository
Acronym: PMMR
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00074547; 1R24DK110492-01 (NIH)
Record Dates: First submitted 2016-09-29; First posted 2016-11-08 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human microbial cell lines, stool and/or DNA and RNA will be collected from participants 10-18 years with a BMI greater than 95th percentile and their healthy siblings.
  Specimens will be collected at 3 time points over a seven month period. Healthy siblings will provide just one blood and stool sample. Samples will be maintained at the Duke Medical Science Research Laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- BMI > 95%: No Intervention
- Healthy Weight Siblings: Control
- Healthy Weight Unrelated: Control

SUMMARY:
The aim of this project is to establish a bio-repository of diverse specimen types to provide investigators access to specimens in order to further research related to metabolism and the microbiome in the pediatric population.

DETAILED DESCRIPTION:
Human microbial cell lines, stool and/or DNA and RNA will be collected from participants 10-18 years with a BMI greater than 95th percentile and their healthy siblings.

Specimens will be collected at 3 time points over a seven month period. Healthy siblings will provide just one blood and stool sample. Samples will be maintained at the Duke Medical Science Research Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Healthy Lifestyles Program at Duke for the care of children with obesity, a sibling of a patient in the Healthy Lifestyles Program, or is a patient at Duke Children's Primary Care.

Exclusion Criteria:

* Pregnant females.

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Samples will be collected upon consent from the patient poplation of the Healthy Lifestyles Program at Duke for the care of children with obesity, a sibling of a patient in the Healthy Lifestyles Program, or is a patient at Duke Children's Primary Care.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2016-09; Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
The measure of abnormal metabolism using a sample biorepository | 5 years
  measures of metabolomics using a sample biorepository

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be shared at investigators discretion following submission of request, receipt of a data transfer agreement and local IRB approval
Time Frame: Data will be available by December 31 2021
Access Criteria: Anonymized data may be shared as investigators discretion following submission of request, receipt of a data transfer agreement and local IRB approval

REFERENCES:
- [Derived] McCann JR, Yang C, Bihlmeyer NA, Tang R, Truong T, An J, Jawahar J, Ilkayeva O, Muehlbauer MJ, Hu Z, Dressman HK, Poppe L, Granek JA, David LA, Shi P, Balikcioglu PG, Shah SH, Armstrong SC, Newgard CB, Seed PC, Rawls JF. Branched chain amino acid metabolism and microbiome in adolescents with obesity during weight loss therapy. medRxiv [Preprint]. 2025 Jun 9:2025.02.03.25321363. doi: 10.1101/2025.02.03.25321363. PMID 39974080